CLINICAL TRIAL: NCT05223036
Title: A Phase IIa, Placebo-Controlled, Randomized Study of Daily Obeticholic Acid (OCA) to Reduce Intestinal Polyp Burden in Familial Adenomatous Polyposis (FAP)
Brief Title: Testing Obeticholic Acid for Familial Adenomatous Polyposis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Partial Clinical Hold
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2022-00341; NCI-2022-00341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0286; 2021-0286 (Other: M D Anderson Cancer Center); MDA20-01-01 (Other: DCP); P30CA016672 (NIH); UG1CA242609 (NIH); NCT05112822 (obsolete NCT alias)
Record Dates: First submitted 2022-02-01; First posted 2022-02-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Attenuated Familial Adenomatous Polyposis; Colorectal Carcinoma; Duodenal Carcinoma; Familial Adenomatous Polyposis
MeSH Terms: conditions — Attenuated familial adenomatous polyposis; Colorectal Neoplasms; Duodenal Neoplasms; Adenomatous Polyposis Coli | interventions — Biopsy; Specimen Handling; Endoscopy, Gastrointestinal; obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (OCA) (Experimental): Patients receive OCA PO QD for 6 months in the absence of unacceptable toxicity. Patients also undergo GI endoscopy with biopsy and collection of blood samples at screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Gastrointestinal Endoscopy; Biological: Obeticholic Acid; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 6 months in the absence of unacceptable toxicity. Patients also undergo GI endoscopy with biopsy and collection of blood samples at screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Gastrointestinal Endoscopy; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Gastrointestinal Endoscopy — Undergo GI endoscopy
  Other Names: Enteroscopy
Biological: Obeticholic Acid — Given PO
  Other Names: INT-747; Ocaliva
  Arms: Arm I (OCA)
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IIa trial investigates if giving obeticholic acid (OCA) is safe and has a beneficial effect on the number of polyps in the small bowel and colon in patients with familial adenomatous polyposis (FAP). FAP is a rare gene defect that increases the risk of developing cancer of the intestines and colon. OCA is a drug similar to a bile acid the body makes. It is fluid made and released by the liver. OCA binds to a receptor in the intestine that is believed to have a positive effect on preventing cancer development. OCA has been effective in treating primary biliary cholangitis (PBC), a liver disease, and is approved by the Food and Drug Administration (FDA) for use at a lower dose (10 mg). There have been studies showing that OCA decreases inflammation and fibrosis. However, it is not yet known whether OCA works on reducing the number of polyps in patients with FAP.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of treatment with OCA versus treatment with placebo on duodenal polyp burden (sum of polyp diameters) in participants with FAP.

SECONDARY OBJECTIVES:

I. To assess the safety profile of treatment with OCA versus placebo in participants with FAP.

II. To evaluate the effect of treatment with OCA versus placebo on rectal and pouch polyp burden (sum of polyp diameters) in participants with FAP.

III. To assess the effect of treatment with OCA versus placebo on polyp burden (absolute number) in the duodenum of participants with FAP.

IV. To assess the effect of treatment with OCA versus placebo on polyp burden (absolute number) in the rectum and rectal pouch of participants with FAP.

V. To evaluate the effect of treatment with OCA versus placebo on serum levels of fibroblast growth factor-19 (FGF19) and 7 alpha-hydroxy-4-cholesten-3-one (7AC4, also known as C4) in participants with FAP.

VI. To determine the effects of treatment with OCA versus placebo on gene expression in duodenal, rectal pouch, and rectal adenomas and uninvolved mucosa in participants with FAP:

VIa. Identify differentially expressed genes between duodenal and colorectal adenomas and uninvolved tissue at baseline and post-intervention for participants who received OCA or placebo; VIb. Quantify the effect of OCA on the expression of downstream targets of FXR in adenomas and uninvolved tissue; VIc. Quantify the effect of OCA on the expression of cancer stem cell markers (e.g. LGR5, ASCL2, LRIG, BMI) and intestinal stem cell markers (e.g. Villin, KRT20, MUC, LYZ) in adenomas and uninvolved tissue.

VII. To evaluate the cell-type specific effects of treatment with OCA versus placebo on gene expression and abundance in duodenal, rectal pouch, and rectal adenomas and uninvolved mucosa in participants with FAP via single-cell transcriptomics.

VIII. To evaluate the effect of treatment with OCA versus placebo on microbiome diversity in duodenal, rectal pouch, and rectal adenomas and uninvolved tissue in participants with FAP.

VIIIa. Compare alpha- and beta-diversity analysis and identify differential abundance in adenomas and uninvolved tissue.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive OCA 25 mg orally (PO) once daily (QD) for 6 months in the absence of unacceptable toxicity. Patients also undergo gastrointestinal (GI) endoscopy with biopsy and collection of blood samples at screening and on study.

ARM II: Patients receive matching placebo PO QD for 6 months in the absence of unacceptable toxicity. Patients also undergo GI endoscopy biopsy and collection of blood samples at screening and on study.

After completion of the study treatment, patients are followed within 14-21 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of phenotypic FAP with disease involvement of the duodenum and rectum as defined by:

  * Genetic diagnosis: APC germline mutation (with or without family history) or obligate carrier
  * Clinical diagnosis: FAP phenotype with > 100 adenomas in large intestine and participant has a family history of FAP
  * Clinical diagnosis: FAP phenotype who are status post colectomy for polyposis, participant has a family history of FAP, and 2 FAP experts agree to the diagnosis
  * Attenuated FAP diagnosis: APC germline mutation required
* Participants must have no evidence of active or recurrent invasive cancer for 6 months prior to screening and must be at least 6 months from any prior cancer-directed treatment (such as surgical resection, chemotherapy, immunotherapy, hormonal therapy or radiation)
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of OCA in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Hemoglobin >= 10 g/dL or hematocrit >= 30%
* Leukocyte count >= 3,500/microliter
* Platelet count >= 100,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Creatinine clearance (calculated if measured is not available) >= 30 mL/min/1.73m^2
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x the institutional upper limit of normal (ULN)
* Total bilirubin =< 1.0 x ULN
* Alkaline phosphatase =< 1.5 x ULN
* Gamma-glutamyl transferase (GGT) =< 1.5 x ULN
* Presence of Spigelman stage II or III duodenal polyposis at screening
* Presence of intact rectum or ileo-rectal anastomosis (IRA) or ileal pouch-anal anastomosis (IPAA) or end ileostomy
* Participants must have a negative test result for human immunodeficiency virus (HIV); if tested within the past 6 months, result will be accepted without repeating the test
* Participants must have negative test for hepatitis C virus (HCV) and B virus (HBV)
* Willing and able to adhere to the prohibitions and restrictions specified in the final approved protocol
* The effects of OCA on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, throughout the duration of study participation, and for at least 6 months after receiving the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Willingness to moderate alcohol intake (consuming no more than 1 or 2 alcoholic drinks per day for women and men, respectively)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior use of study drug
* Duodenal or rectal/pouch polyp burden that is not quantifiable
* Histologically-confirmed high-grade dysplasia or cancer on biopsy at screening
* Individuals with active, known or suspected chronic liver disease including cirrhosis, nonalcoholic steatohepatitis (NASH) with liver fibrosis, NASH with cirrhosis, primary sclerosing cholangitis, biliary atresia
* Individuals with acute cholecystitis (defined by a syndrome of right upper quadrant pain, fever, and leukocytosis associated with gallbladder inflammation)
* Individuals with a history of pancreatitis or presence of pancreatic abnormalities suggestive of increased risk of pancreatitis
* Individuals with hepatic steatosis and velocity > 1.7 meters/second (m/s) as determined by liver ultrasound elastography
* Individuals with hyperlipidemia not well controlled with the use of pharmacotherapy and/or dietary modifications
* History of severe, progressive, or uncontrolled renal, genitourinary, hepatic, hematologic, endocrine, cardiac, vascular, pulmonary, rheumatologic, neurologic, psychiatric, or metabolic disturbances, or signs and symptoms thereof
* Pregnant, breast-feeding, or women of childbearing potential unwilling to use a reliable contraceptive method. Pregnant women are excluded from this study because OCA is an agent with unknown effects on the developing human fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OCA, breastfeeding should be discontinued if the mother is treated with OCA
* Known hypersensitivity, allergies, or intolerance to the study drug or compounds of similar chemical or biologic composition
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures
* Participants may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Individuals with active and untreated hepatitis C virus (HCV) and/or or hepatitis B virus (HBV) infection
* Individuals with HIV infection are eligible for participation if:

  * CD4+ count >= 300/uL
  * Viral load is undetectable
  * Receiving highly active antiretroviral therapy (HAART) without known or suspected drug interactions with OCA
  * Consultation with the participant's infectious disease specialist may be obtained
* Individuals taking the drugs listed below may not be randomized unless they are willing to stop the medications (and possibly change to alternative non-excluded medications to treat the same conditions) no less than 5 half-lives days prior to starting OCA or placebo on this study. Consultation with the participant's primary care provider may be obtained but is not required. The use of the following drugs or drug classes is prohibited during OCA/placebo treatment:

  * Investigational agents
  * Bile acid sequestrants (bile acid binding resins): cholestyramine, colestipol, or colesevelam
  * Bile salt efflux pump (BSEP) inhibitors
  * Clozapine
  * Theophylline derivatives
  * Tizanidine
  * Warfarin
  * Hepatotoxic drugs such as amiodarone, sodium valproate, certain herbal/dietary supplements, and long-term doxycycline or tetracycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-02-21 (Estimated)

PRIMARY OUTCOMES:
Percentage change in duodenal polyp burden | Baseline to 6 months
  Change from baseline will be summarized by treatment arm. The difference in change from baseline between active treatment arms and the placebo arm will also be summarized.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 21 days after completion of treatment
  Will summarize adverse events for each group by grade and study drug attribution using descriptive statistics.
Absolute differences in the levels of serum FGF19 and C4 | Baseline to 6 months
  Differences in the median serum levels of FGF19 and C4 between treatment arms will be compared.
Percentage change in the number of duodenal polyps | Baseline to 6 months
  Will use parametric models to evaluate the absolute and/or relative changes from baseline of these measures between obeticholic acid (OCA) and placebo groups.
Percentage change in the number of colorectal, rectal/pouch polyps | Baseline to 6 months
  Will use parametric models to evaluate the absolute and/or relative changes from baseline of these measures between OCA and placebo groups.
Percentage change in colorectal, rectal/pouch polyp burden | Baseline to 6 months
  Will use parametric models to evaluate the absolute and/or relative changes from baseline of these measures between OCA and placebo groups.
Changes in gene expression (messenger ribonucleic acid) profiles of adenomas and normal mucosa | Baseline to 6 months
  Will apply methods such as the beta-uniform mixture (BUM) model, the Wilcoxon rank-sum test with empirical Bayes, and the significance analysis of microarrays (SAM) to control the first degree relative (FDR).
Changes in the microbiome of adenomas and normal mucosa | Baseline to 6 months
  Will apply methods such as the BUM model, the Wilcoxon rank-sum test with empirical Bayes, and the SAM to control the FDR.
Future candidate biomarkers measured by genomic and transcriptomic platforms in residual tissue biopsies of adenomas and normal mucosa | At 6 months
  Will apply methods such as the BUM model, the Wilcoxon rank-sum test with empirical Bayes, and the SAM to control the FDR.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar-Sanchez, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - M D Anderson Cancer Center, Houston, Texas
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm